CLINICAL TRIAL: NCT01378715
Title: Rosuvastatin Pre-Treatment Influences the Risk of Percutaneous Coronary Intervention Study (TIPS-3)
Brief Title: Rosuvastatin Pre-Treatment Influences the Risk of Coronary Intervention Study
Acronym: TIPS-3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Prof. Jan Trka, MD, PhD, 2nd Medical School of Charles University and University Hospital Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-134/10
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; statins; periprocedural myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator): Patients with coronary artery disease referred for coronary angiography and subsequently PCI will be enrolled and randomized to pre-treatment with rosuvastatin (20mg 12 hours prior + 20mg immediately prior PCI).
  Interventions: Drug: Rosuvastatin
- Control (No Intervention): Patients with coronary artery disease referred for coronary angiography and subsequently PCI will be enrolled and randomized to no-pretreatment with rosuvastatin.

INTERVENTIONS:
Drug: Rosuvastatin — Patients with coronary artery disease referred for coronary angiography and subsequently PCI will be enrolled and randomized to pre-treatment with rosuvastatin (20mg 12 hours prior + 20mg immediately prior PCI).
  Other Names: Rosucard (Zentiva, Czech Republic)
  Arms: Rosuvastatin

SUMMARY:
The aim of this study is to determine whether a pre-treatment with high-dose statin (one day prior and just before intervention, rosuvastatin 20mg/day) has a positive impact on the occurrence of periprocedural myocardial infarction during percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The aim of this study is to attest whether a short-term treatment with high-dose statin (one day prior and before intervention, rosuvastatin 20mg/day) can have a positive impact over the occurrence of periprocedural myocardial infarction during percutaneous coronary intervention (PCI). Patients with stable or unstable (with negative troponin) angina pectoris receiving statins (or not, except rosuvastatin 40mg a day) therapy referred for coronary angiography and subsequently PCI will be enrolled and randomized (ratio 1:1) to pre-treatment with rosuvastatin (20mg 12 hours prior + 20mg immediately before PCI - Rosuvastatin group), or immediate PCI (control group). Serum concentration of troponin I will be measured prior to, 12 hours and 24 hours after PCI.

Power of study (200 vs 200 pts; p1 = 0.2; p2 = 0.33; alfa = 0.05, n1 = 200, n2 = 200; power 0.84).

The primary end-point will be the TnI concentration ≥ 1.5 times the ULN. The secondary end-point witl be the TnI concentration ≥ 3 times ULN.

The Cox regression model will be used to identify the predictors of primary end-points (age, diabetes, smoking, symptomatic peripheral artery disease, statin pre-treatment, level of total cholesterol, pre-treatment with clopidogrel, multi-vessel disease, unstable angina, hs-CRP, therapy with beta-blockers, treatment of complex coronary lesion).

The patient included shall fulfill all the criteria: 1) significant coronary artery stenosis or occlusion indicated for percutaneous coronary intervention and 2) signed informed consent.

The criteria excluding the inclusion in the study are: 1) positive troponin I (≥ 1 ULN), 2) previous inclusion in this study, 3) renal insufficiency, 4) chronic treatment with rosuvastatin 40mg or more, and 5) disagreement to be included in this study.

This study will be multicenter. The Motol University Hospital will participate as the project coordinator.

ELIGIBILITY:
Inclusion Criteria:

* significant coronary artery stenosis or occlusion indicated for percutaneous coronary intervention
* signed informed consent

Exclusion Criteria:

* positive troponin I (≥ 1 ULN)
* previous inclusion in this study
* renal insufficiency (creatinine ≥ 200 umol/l)
* chronic treatment with rosuvastatin 40mg or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
periprocedural myocardial infarction during percutaneous coronary intervention | 24 hours after PCI
  TnI concentration ≥ 1.5 times the ULN

SECONDARY OUTCOMES:
periprocedural myocardial infarction during percutaneous coronary intervention | 24 hours after PCI
  TnI concentration ≥ 3 times ULN

CONTACTS AND LOCATIONS:
Overall Officials: Josef Veselka, Prof., MD, Study Chair — Dpt. of Cardiology, 2nd Medical School of Charles Universty and University Hospital Motol; David Zemanek, MD, Study Director — Dpt. of Cardiology, 2nd Medical School of Charles Universty and University Hospital Motol
Locations (4):
- Czechia (3):
  - 1st Medical Dept., Faculty of Medicine in Plzen, Charles University in Prague, University Hospital Plzen, Pilsen
  - Dpt. of Cardiology, 2nd Medical School of Charles Universty and University Hospital Motol, Prague
  - Dpt. of Cardiology, Hospital Podlesi, Třinec
- Eastern Slovakia Institute of Cardiovascular Diseases, Košice, Slovakia